CLINICAL TRIAL: NCT02037971
Title: Effectiveness of Exercise Training in Improving Sleep in Patients With Systemic Lupus Erythematosus: A Controlled Randomized Trial.
Brief Title: Aerobic Exercise on Improving Sleep in Systemic Lupus Erythematosus.
Acronym: EFEXO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Lilian K C Reis, Principal Investigator, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 03315312.8.0000.5505
Record Dates: First submitted 2013-03-24; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-05

CONDITIONS: Systemic Lupus Erythematosus; Sleep Disorders
Keywords: Systemic Lupus Erythematosus; Lupus; Sleep disorders; Sleep disturbed; Physical exercise; Aerobic exercise
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sleep Wake Disorders; Parasomnias; Motor Activity | interventions — Exercise; Physical Conditioning, Human; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (Experimental): Subjects will follow one defined exercise process, according their cardiopulmonary exercise test, during 16 weeks, two times per a week.
  Interventions: Procedure: Aerobic Exercise
- Control Group (Experimental): A non-exercise group will receive regular educational information relating to their condition.
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: Aerobic Exercise — From 1st week up to and including 4th week, subjects will do: 5 minutes warm-up, then 15-30 minutes low to moderate (55-65% VO2) exercise, then 15 minutes stretching. From 5th week up to and including 16th week, subjects will do: 5 minutes warm-up, then intermittent training for between 30-40 minutes, then 10 minutes stretching.
  Other Names: Physical activity; Physical training
  Arms: Aerobic Exercise
Other: Control Group — The control group will have monthly meetings to learn about: good sleep habits, Systemic Lupus Erythematosus (their disease) and general good health.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine the effectiveness of exercise training on improving sleep in patients with systemic lupus erythematosus.

DETAILED DESCRIPTION:
This study will test the effectiveness of aerobic exercise on improving sleep in patients with systemic lupus erythematosus. The subjects will do treadmill 2 times per week, from 15-20 min. with low to moderate(55-65% maxCF) intensity exercise, so 30 min. until 4ª week. From the 5ª to 8ª week they will be able to make greater efforts to 35-40 min. totalizing 16 weeks. The control group will not do exercise and will receive education class about disease, health, sleep, 1 time per month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Lupus Erythematosus (SLE) according American College of Rheumatology (ACR) Criteria revised in 1997;
* Pittsburgh sleep quality index (PSQI) ≥ 5;
* Free and Clarified Consent Term signature.

Exclusion Criteria:

* Patients who have other rheumatologic diseases (rheumatoid arthritis, sjogren syndrome, fibromyalgia, ankylosis spondylitis), excerpt mild osteoarthritis;
* Systemic Lupus Erythematosus Disease Assessment Index (SLEDAI) > 8;
* Untreated diseases: Hypertension, diabetes mellitus (DM), dyslipidemia, thyroid dysfunction, cardiorespiratory diseases, malignancies;
* Patients who do not accept the study rules as time and/or follow-up exercise program time proposed;
* Suspected or pregnancy confirmation;

  * Patients who are taking sleeping medication;
* Patients who won´t sign the Free and Clarified Consent Term informed;
* Patients engaged in physical activity (defined as previously sedentary individuals, or that which do not perform any type of regular physical activity at least six months);

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | 16 weeks
  Sleep efficiency will be evaluate with actigraph. The subject will use it for 15 days before the period of exercise, 15 days at the start of the period of exercise, and then 15 last days in the period of exercise.
  Complementing the information collected by the device, the patient will complete a sleep diary, with schedules of activities such as: time they go to bed, time they fall asleep, time they get up, times they remove the device (which is not waterproof), times they replace the device, and times they wake up from naps.
Sleep quality | 16 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire that includes 21 items that assess the quality of sleep during a one-month period.
  The subject will be asked it, before, during and after the period of exercise. The questionnaire is divided into seven components: subjective sleep quality, sleep latency, sleep duration, sleep effectiveness, sleep disorder, use of sleep medication, and daytime dysfunction.
  On the PSQI a score ≥ 5 indicates poor quality of sleep, and ≤ 4 indicates good quality of sleep.

SECONDARY OUTCOMES:
Pain assessment | 16 weeks
  Subjects' pain will be assessed utilizing the Visual Analogue Scale (VAS) which consists of a numeric range from 1 to 10, where 1 represents light pain and 10 represents intense pain.
Disease activity assessment | 16 weeks
  Subjects' disease activity will be evaluated using SLEDAI, a modification of the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI). It is a list of 24 clinical and laboratory items which assess and quantify disease activity. A subject's score has to be ≤ 8 to be considered for the study.
Quality of life assessment | 16 weeks
  Subjects' health will be evaluated utilizing the questionnaire 'Short Form (36) Health Survey' (SF-36).
Restless Legs Syndrome gravity assessment | 16 weeks
  Subjects' Restless Legs Syndrome (RLS) gravity will be assessed using the International Restless Legs Syndrome Rating Scale. It consists in 10 questions that evaluate the severity of symptoms and impact of the disease on daily life activities.
Fatigue assessment | 16 weeks
  Subjects' fatigue will be evaluated using the Fatigue Severity Scale (FSS) which consists of 9 questions and a numeric range from 1 to 7, where 1 represents minimum severity and 7 represents maximum severity.
Fatigue assessment | 16 weeks
  Subjects' fatigue will be evaluated using the Visual Analogue Scale for overall fatigue (VAS-fatigue) which consists of a numeric range from 1 to 10, where 1 represents light fatigue and 10 represents intense fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian KC Reis, Study Chair — Federal University of São Paulo UNIFESP; Virginia FM Trevisani, Principal Investigator — Federal University of São Paulo
Locations (1):
- Psychobiology and Exercise Studies Centre, São Paulo, São Paulo, Brazil